CLINICAL TRIAL: NCT01480622
Title: An Open-label Single and Repeat Dose Study to Investigate the Pharmacokinetic Profiles of Tenofovir Disoproxil Fumarate 300 mg in Healthy Chinese Subjects
Brief Title: Pharmacokinetic (PK) Profiles of Tenofovir Disoproxil Fumarate (TDF) 300 mg in Healthy Chinese Subjects
Acronym: PK of TDF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115515
Record Dates: First submitted 2011-11-17; First posted 2011-11-29 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis B, Chronic
Keywords: healthy subjects; Tenofovir disoproxil fumarate; hepatitis; pharmacokinetics
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TDF tablets (Experimental): Tenofovir disoproxil fumarate tablets
  Interventions: Drug: TDF tablets

INTERVENTIONS:
Drug: TDF tablets — White, almond-shaped, film-coated tablets, one side with the markings "GILEAD" and "4331"

SUMMARY:
This study will evaluate the pharmacokinetic profile of tenofovir disoproxil fumarate (TDF) 300 mg in Chinese subjects to support the registration of this compound in the People's Republic of China. This will be an open-label, single group, single and repeat dose study without placebo in healthy male and female subjects. Pharmacokinetic sampling to enable measurement of plasma concentrations of tenofovir will be conducted over a 60-h period after the single dose and at steady state. The duration of the study will be approximately 7 weeks from screening to follow-up.

DETAILED DESCRIPTION:
This will be an open-label, single group, single and repeat dose study with no placebo control in healthy Chinese subjects conducted at a single centre. The study will include a screening visit, single and repeat dose sessions and a follow-up contact.

The screening visit will be conducted up to 28 days prior to the first dose of treatment period 1. Screening assessments will occur as indicated in the Time and Events Table.

Subjects who meet the inclusion/exclusion criteria will be admitted to the study centre on Day -1 to undergo baseline procedures before the single dose session. Study medication will be administered the following morning (Day 1) for the single dose phase. Subjects will be required to fast for at least 8 h (overnight) prior to dosing until 4 h after dosing. Pharmacokinetic samples will be taken until Day 3.

The repeat dose session will begin on Day 4. Subjects will receive a once daily dose of TDF 300 mg in a fasted state each morning for 7 days. Subjects will be required to fast for at least 8 h (overnight) prior to dosing on Day 8 and Day 9, and for at least 8 h (overnight) prior to dosing until 4 h after dosing on Day 10. A trough pharmacokinetic sample will be collected before dosing on Day 8, Day 9 and a series of samples will be taken from Day 10 to Day 12.

Subjects will remain in-house from the evening before dosing (Day -1) until after the final pharmacokinetic sample has been collected on Day 12 and the final safety assessment completed on Day 13. Then subjects will be discharged from the study centre at the Investigator's discretion.

Subjects completing the dosing sessions will not be required to visit the study centre for a follow-up visit, unless the Investigator determines that it is necessary for safety or other reasons. All subjects will receive a follow-up contact by telephone or visit 7 days after the last dosing to collect any information on concomitant medication taken and AEs experienced since the last visit.

The total duration of each subject's participation, from screening to follow-up contact, will be approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by a responsible and experienced physician
* Male or female between 18 and 45 years of age
* Body weight >50 kg (110 lbs) for males or >45 kg (100 lbs) for females, and body mass index (BMI) between 19.0 and 24.0 kg/m2

Exclusion Criteria:

* Positive result for hepatitis B, hepatitis C or HIV at screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* Positive urine drug screen and breath alcohol test at screening or prior to dosing
* Lactating females

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12-05 (Actual); Primary Completion 2011-12-30 (Actual); Study Completion 2011-12-30 (Actual)

PRIMARY OUTCOMES:
area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC(0-t)) | up to 60 hours after single dose
  AUC(0-t) of single dose
area under the concentration-time curve during steady state (AUC(0-τ)) | up to 60 hours after repeat dose
  AUC(0-τ) during steady state

SECONDARY OUTCOMES:
adverse events (AEs) | up to 20 days, from the first dose until the follow-up contact
  AEs accur during the study
vital signs | day 1 pre-dose, day 2, day 3, day 10 pre-dose, day 11, day 12 and day 13 prior to discharge from hospital
  blood pressure, pulse rate, respiratory rate and temperature
lab assessment | day 13, prior to discharge from hospital
  Haematology, Clinical Chemistry and Routine Urinalysis
12-lead electrocardiogram (ECG) parameters | day 13, prior to discharge from hospital
  the heart rate and measures PR, QRS, QT and QTc intervals. All ECGs must be evaluated for safety by a qualified physician.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

REFERENCES:
- [Derived] Hu CY, Liu YM, Liu Y, Chen Q, Wang W, Wu K, Dong J, Li J, Jia JY, Lu C, Sun SX, Yu C, Li X. Pharmacokinetics and tolerability of Tenofovir disoproxil fumarate 300 mg once daily: an open-label, single- and multiple-dose study in healthy Chinese subjects. Clin Ther. 2013 Dec;35(12):1884-9. doi: 10.1016/j.clinthera.2013.09.020. Epub 2013 Oct 19. PMID 24148552
- See also: Results for study 115515 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115515?search=study&search_terms=115515#rs